CLINICAL TRIAL: NCT00363324
Title: Effects of Autologous Bone Marrow Celss on Acute ST-Elevation Myocardial Infarction
Brief Title: Bone Marrow Cells in Myocardial Infarction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Oulu (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 82/04
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2008-01-09 (Estimated); Status verified 2007-12

CONDITIONS: Acute Myocardial Infarction
Keywords: stem cell; acute myocardial infarction

INTERVENTIONS:
Procedure: intracoronary injection of bone marrow cells

SUMMARY:
This study is aimed to assess the effect of bone marrow cells on arrhythmia risk variables in patients with a acute myocardial infarction.

DETAILED DESCRIPTION:
This is a randomized, double-blinded study, where patients treated with thrombolytic therapy for acute myocardial infarction are randomized to receive bone-marrow derived stem cells or sham-infusion at the time percutaneous coronary intervention of the target vessel. The end-points are many arrhythmia risk variables, suchs as heart rate variability, T-wave alternans and many ECG variables as well as systolic and diastolic left ventricular function.

ELIGIBILITY:
Inclusion Criteria:

* Acute ST-elevation myocardial infarction treated with thrombolytic therapy

Exclusion Criteria:

* Indication for rescue PCI, severe clinical heart failure, age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Arrhythmia risk variables
left ventricular function
restenosis assessed by IVUS

SECONDARY OUTCOMES:
exercise tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Heikki V Huikuri, Professor, Principal Investigator — University of Oulu
Locations (1):
- University of Oulu, Oulu, Finland

REFERENCES:
- [Derived] Miettinen JA, Salonen RJ, Niemela M, Kervinen K, Saily M, Koistinen P, Savolainen ER, Ukkonen H, Pietila M, Airaksinen KE, Knuuti J, Makikallio TH, Huikuri HV, Ylitalo KV. Effects of intracoronary infusion of bone marrow-derived stem cells on pulmonary artery pressure and diastolic function after myocardial infarction. Int J Cardiol. 2010 Dec 3;145(3):631-3. doi: 10.1016/j.ijcard.2010.09.064. Epub 2010 Oct 20. No abstract available. PMID 20961630
- [Derived] Miettinen JA, Ylitalo K, Hedberg P, Jokelainen J, Kervinen K, Niemela M, Saily M, Koistinen P, Savolainen ER, Ukkonen H, Pietila M, Airaksinen KE, Knuuti J, Vuolteenaho O, Makikallio TH, Huikuri HV. Determinants of functional recovery after myocardial infarction of patients treated with bone marrow-derived stem cells after thrombolytic therapy. Heart. 2010 Mar;96(5):362-7. doi: 10.1136/hrt.2009.171694. Epub 2009 Nov 11. PMID 19910293
- [Derived] Huikuri HV, Kervinen K, Niemela M, Ylitalo K, Saily M, Koistinen P, Savolainen ER, Ukkonen H, Pietila M, Airaksinen JK, Knuuti J, Makikallio TH; FINCELL Investigators. Effects of intracoronary injection of mononuclear bone marrow cells on left ventricular function, arrhythmia risk profile, and restenosis after thrombolytic therapy of acute myocardial infarction. Eur Heart J. 2008 Nov;29(22):2723-32. doi: 10.1093/eurheartj/ehn436. Epub 2008 Oct 9. PMID 18845667